CLINICAL TRIAL: NCT01629953
Title: Assessing Supported Employment With Veterans With Felony Convictions and MI or SA
Brief Title: Assessing Supported Employment With Veterans With Felony Convictions and Mental Illness or Substance Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7635-R
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Results first posted 2018-05-22 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Employment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Based Vocational Rehabilitation (Active Comparator): Group vocational intervention
  Interventions: Other: Group vocational intervention
- Supported Employment Condition (Experimental): Group vocational intervention + supported employment
  Interventions: Other: Supported Employment Condition

INTERVENTIONS:
Other: Group vocational intervention — Group based manualized vocational rehabilitation
  Arms: Group Based Vocational Rehabilitation
Other: Supported Employment Condition — Veterans in this condition will receive a proven group based manualized vocational rehabilitation intervention
  Arms: Supported Employment Condition

SUMMARY:
This study continues to develop and refine best practices in the delivery of vocational services to veterans with histories of felony convictions and mental health/substance abuse difficulties. There are currently over 225,000 incarcerated veterans and it is estimated 64,000 veterans are released from prisons annually. These veterans encounter significant difficulties in finding employment due to stigma, intrapersonal difficulties, and out-dated work skills. Additionally these veterans are more likely to be homeless than other population., Previous work has found that manual based, vocational groups led by trained vocational staff led to quicker employment compared to traditional vocational services and manual based self studies. To attempt to improve on previous results, this study adds principles and components of supported employment including ongoing follow-up, treatment team coordination, and community based assistance.

ELIGIBILITY:
Inclusion Criteria:

* history of at least one felony conviction
* diagnosis of a mental illness including substance use disorders

Exclusion Criteria:

* dementia
* active psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P. LePage, PhD, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (1):
- VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group Based Vocational Rehabilitation | Supported Employment Condition
Started | 65 | 75
Completed | 52 | 60
Not Completed | 13 | 15
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 10 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Based Vocational Rehabilitation | Supported Employment Condition | Total
Number analyzed (Participants) | 52 | 60 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 60 | 111
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (5.4) | 51.5 (5.8) | 52.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 52 | 59 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  racial or ethnic minority | 39 | 43 | 82
Region of Enrollment [Number; unit: participants]
  United States | 52 | 60 | 112

OUTCOME MEASURES:

1. Primary Outcome: Employment
Description: Number of veterans finding work within 6 months
Time Frame: within 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group Based Vocational Rehabilitation | Supported Employment Condition
Number analyzed (Participants) | 38 | 46
Participants | 8 | 21

2. Primary Outcome: Total Employment
Description: Total amount employed over 1 year follow-up period
Time Frame: 1 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group Based Vocational Rehabilitation | Supported Employment Condition
Number analyzed (Participants) | 52 | 60
Participants | 19 | 34

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group Based Vocational Rehabilitation | Supported Employment Condition
All-Cause Mortality (participants affected / at risk) | 1/52 | 5/60
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/60
Other Adverse Events (participants affected / at risk) | 0/52 | 0/60

LIMITATIONS AND CAVEATS:
Continual follow-up was difficult and though all 112 had post data recorded, not all Veterans had monthly updates. This may have led to some loss of specific start dates for employment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No